CLINICAL TRIAL: NCT07098091
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of Single and Multiple Doses of YD0293 Tablets in Healthy Subjects
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of YD0293 in Healthy Subjects
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Yidian Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Shanghai Huilun Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PY-YD0293-I-01
Record Dates: First submitted 2025-07-16; First posted 2025-08-01 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-05

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YD0293 (Experimental): Single dose ascending(SAD): participants will be randomized to receive a single dose of YD0293, dose ascending will be conducted sequentially from the low-dose cohort to the high-dose cohort.
  Multiple ascending dose(MAD): participants will be randomized to receive muliple doses of YD0293, dose ascending will be conducted sequentially from the low-dose cohort to the high-dose cohort.
  Food effect(FE): participants will be randomized to group A or group B, to evaluate different fed conditions on the PK of YD0293.
  Interventions: Drug: YD0293
- YD0293 placebo (Placebo Comparator): Single dose ascending(SAD): participants will be randomized to receive a single dose of placebo, dose ascending will be conducted sequentially from the low-dose cohort to the high-dose cohort.
  Multiple ascending dose(MAD): participants will be randomized to receive muliple doses of placebo, dose ascending will be conducted sequentially from the low-dose cohort to the high-dose cohort.
  Food effect(FE): participants will be randomized to group A or group B, to evaluate different fed conditions on the PK of YD0293.
  Interventions: Drug: YD0293 placebo

INTERVENTIONS:
Drug: YD0293 — YD0293 tablet for oral administration
  Arms: YD0293
Drug: YD0293 placebo — YD0293 placebo tablet for oral administration
  Arms: YD0293 placebo

SUMMARY:
This study is a single-center, single- and multiple-dose escalating study with a food-effect component, designed to evaluate the safety, tolerability, and pharmacokinetic (PK) characteristics of YD0293 tablets following a single oral dose in healthy subjects, as well as the effect of food on PK parameters and the potential effect on the QT interval. The study also aims to assess the safety, tolerability, and PK profile of YD0293 tablets following multiple oral doses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, both male and female, in each group;
2. 18 years old< = age< = 45 years old;
3. The weight of men shall not be less than 50kg, and the weight of women shall not be less than 45kg. Body mass index (BMI) = weight (kg) / height ^2 (m^2), 19.0kg/m2< = body mass index (BMI) < = 26.0 kg/m^2;
4. During the screening period, those who have undergone vital signs, physical examination, blood routine, blood biochemistry, coagulation function, urine routine, virological examination, chest X-ray, B-ultrasound and blood pregnancy (female), and the results show no abnormality or abnormality without clinical significance;
5. The results of the 12-lead ECG during the screening period are consistent with normal cardiac conduction and function, including: Sinus rhythm, 50< = heart rate < = 100 bpm; b. QT interval (QTcF) corrected using Fridericia method <=450 ms; c. QRS<=120 ms; d. PR interval <=210 ms; e. The ECG morphology is normal, and there are no clinically significant changes as judged by the investigator.
6. The subject agrees to have no fertility plan and voluntarily take effective contraceptive measures during the trial period and within 3 months after the last dose;
7. The subjects fully understand the purpose, nature, methods and possible adverse events of the trial, voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding females;
2. History of chronic diseases or clinical abnormalities that need to be excluded, including but not limited to disorders of the central nervous system, cardiovascular system, kidneys, liver, gastrointestinal tract, respiratory system, hematologic system, metabolic disorders, and musculoskeletal system, or any other physiological condition that could interfere with study results;
3. Active infectious disease requiring antimicrobial treatment at screening;
4. Undergone surgery within 3 months prior to screening and not fully recovered, as judged by the investigator;
5. Previous or current diagnosis of functional dipeptidyl peptidase-1 (DPP1) deficiency leading to periodontitis or palmoplantar keratoderma, with current signs of gingivitis/periodontitis or a history of palm or sole hyperkeratosis or erythema;
6. Confirmed clinically significant allergic reactions (e.g., to food, any component of the investigational drug or placebo, atopic reactions, asthma attacks), which the investigator believes would interfere with the subject's participation in the trial;
7. Clinically relevant immunosuppressive diseases (including but not limited to immunodeficiency disorders);
8. Abnormal liver function test results (e.g., AST, ALT, GGT) deemed clinically significant by the investigator;
9. Abnormal creatine kinase MB (CK-MB) levels deemed clinically significant by the investigator;
10. Participation in another drug or medical device clinical trial within 3 months prior to screening;
11. Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus IgG antibody, HIV antibodies and p24 antigen, or anti-treponemal antibody at screening, and considered clinically significant by the investigator;
12. Presence of tattoos or scars on any part of the skin that would affect safety assessments, as judged by the investigator;
13. Received vaccination within 1 month prior to screening or during the screening period;
14. History of blood donation within 3 months prior to screening, or plans to donate blood or blood components during the study period, or total blood loss >= 200 mL due to bleeding (excluding menstrual bleeding);
15. Taken any medication within 2 weeks prior to dosing, including strong inhibitors or inducers of CYP3A4 or CYP2D6, traditional Chinese medicine, weight-loss drugs, or supplements;
16. Consumed excessive amounts of tea, coffee, or caffeine-containing beverages (more than 8 cups per day, 1 cup = 250 mL) within 3 months prior to screening;
17. Regular alcohol consumption (more than 14 units per week; 1 unit = 360 mL beer or 45 mL of 40% spirits or 150 mL wine) within 6 months prior to screening or during the screening period, and unable to abstain from alcohol during the trial;
18. Smoked >= 5 cigarettes per day within 6 months prior to screening, or unable to stop using tobacco products during the trial;
19. Unable to refrain from smoking, consuming alcohol (or alcoholic beverages), tea, or coffee from 48 hours before dosing until the last blood draw;
20. Consumed large quantities of grapefruit, pomelo, star fruit, mango, or dragon fruit drinks or foods within 14 days prior to screening or within 48 hours before the first dose;
21. History of drug abuse within 5 years prior to screening or positive urine drug screen (morphine, THC, methamphetamine, MDMA, ketamine);
22. Engaged in strenuous exercise within 1 week prior to dosing, or unable to stop strenuous exercise during the trial;
23. History of torsades de pointes or other risk factors, or family history of short QT syndrome, long QT syndrome, unexplained sudden death or drowning under age 40, or SIDS in first-degree relatives (biological parents, siblings, or children), or presence of implanted pacemaker or ICD;
24. Applicable only to FE studies: Special dietary requirements that prevent adherence to a standardized diet or difficulty swallowing;
25. Unable to tolerate venipuncture or difficult with blood sampling;
26. Any other condition deemed unsuitable for participation by the investigator;
27. Subject requests withdrawal from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of YD0293 in healthy participants | Single ascending dose(SAD): day1 to day15; Multiple ascending dose(MAD): day1 to day39; Food effect(FE): day1 to day21
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
To assess the pharmacokinetic parameters of YD0293 in healthy participants | Single ascending dose(SAD): day1 to day5; Multiple ascending dose(MAD): day1 to day32; Food effect(FE): day1 to day11
  Time to reach maximum concentration (Tmax)
To assess the pharmacokinetic parameters of YD0293 in healthy participants | Single ascending dose(SAD): day1 to day5; Multiple ascending dose(MAD): day1 to day32; Food effect(FE): day1 to day11
  Maximum concentration (Cmax)
To assess the pharmacokinetic parameters of YD0293 in healthy participants | Single ascending dose(SAD): day1 to day5; Multiple ascending dose(MAD): day1 to day32; Food effect(FE): day1 to day11
  Area under the plasma concentration-time curve from time 0 to last time of quantifiable concentration (AUC0-t)
To assess the pharmacokinetic parameters of YD0293 in healthy participants | Single ascending dose(SAD): day1 to day5; Multiple ascending dose(MAD): day1 to day32; Food effect(FE): day1 to day11
  Elimination half time (T1/2)
To assess the changes in QT/QTc intervals following a single oral dose of YD0293 tablets | Single ascending dose(SAD): day1 to day2
To assess the pharmacodynamic characteristic of YD0293 in healthy participants | Multiple ascending dose(MAD): day1 to day32
  Change in active neutrophil elastase concentrations in blood after multiple oral doses of YD0293 from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jie Pan, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China